CLINICAL TRIAL: NCT06349863
Title: Variation in Cholecystitis Treatment and Outcome in the Netherlands; a Nation-wide Cohort Study
Brief Title: Dutch Cholecystitis Snapshot Study
Acronym: Dutch CHESS
Status: Recruiting | Type: Observational
Sponsor: St. Antonius Hospital (Other)
Collaborators: St. Antonius Onderzoeksfonds (Unknown); Dutch Snapshot Research Group (Unknown); Nederlandse Leverpatientenvereniging (Unknown)
Responsible Party: Principal Investigator, Teus Weijs, Principal Investigator, St. Antonius Hospital
Other Study IDs: W23.225
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Cholecystitis; Cholecystitis; Gallstone; Cholecystitis; Choledocholithiasis
MeSH Terms: conditions — Cholecystitis; Gallstones; Choledocholithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Cholecystitis is treated by in various types of hospitals by different specialists, and treatment strategy is influenced by logistical and medical reasons and personal preference. This may significantly impact hospital stay and other outcomes.

Purpose: To determine the variation in treatment of cholecystitis in the Netherlands and its impact on outcome.

Methods: Nation-wide cohort study of all patients diagnosed and treated for cholecystitis during a 6 month period. The primary outcome will be the proportion of patients with an acute cholecystitis in which the guideline is followed. This group will be compared to those in which the guideline is not followed, focussing on total hospital stay and complications. Secondary aims are to determine: factors related to guideline compliance; the best method of cystic duct closure; the best treatment strategy for a >7-day existing cholecystitis; factors predictive for concomitant common bile duct stones; strategies following gallbladder drainage. Multivariable analysis and propensity score matching will be used when appropriate for the etiological study aims. The TRIPOD guideline for prediction modelling will be used for the predictive study aims. Hospitals will receive their own results, set out against the national average and best practices, thereafter subsequent changes in hospital practice will be recorded.

Conclusion: This study will determine the variation in treatment of cholecystitis in the Netherlands and its impact on clinical outcome. Its results will serve as an important incentive to create optimal, uniform cholecystitis treatment in the Netherlands.

ELIGIBILITY:
All patients >18 years with a calculous cholecystitis as primary reason for their hospital admittance. Location of diagnosis may the emergency department, the ward during admittance for diagnostics, or during diagnostic laparoscopy. Cholecystitis is defined according to the TG18 diagnostic criteria for a definitive diagnosis of cholecystitis: A. Local signs of inflammation (Murphy's sign and or RUQ mass/pain/tenderness) + B. Systemic signs of inflammation (Fever, elevated CRP and/or elevated WBC count) + C. Imaging findings characteristic of acute cholecystitis. Patients with a suspected diagnosis (one item in A + one item in B + C), of which the diagnosis is confirmed by peroperative findings, are also included. Patients will be identified by a local study investigator, e.g. a surgeon or surgeon in training.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is descibed under in/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Total hospital stay | First six months following diagnosis
  Median (IQR) or mean (+/-SD) hospital stay in days for patients diagnosed with calculous cholecystitis for the cholecystitis or new complications related to their gallstones following the initial cholecystitis episode, this also includes admission for complications of treatments received. This is the primary outcome for the primary comparison: patients with a 0-7 day cholecystitis receiving early cholecystectomy conform the guidelines versus patients with a 0-7 day cholecystitis who receive alternative treatments.

CONTACTS AND LOCATIONS:
Locations (1):
- Heelkunde, Nieuwegein, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Maasakkers MHG, Weijs TJ, Goense L, van Lienden KP, van Duijvendijk P, Verdonk RC, Boerma D. Uncovering variation in cholecystitis treatment: protocol and statistical analysis plan for a nationwide observational study - the Dutch Cholecystitis Snapshot Study (Dutch CHESS). BMJ Open. 2025 May 13;15(5):e093821. doi: 10.1136/bmjopen-2024-093821. PMID 40360397